CLINICAL TRIAL: NCT01495091
Title: Markers of Coronary Artery Disease During Exercise Testing
Acronym: CADENCE
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Arnljot Flaa, Dr, Oslo University Hospital
Other Study IDs: 2011/1938 (REK)
Record Dates: First submitted 2011-12-09; First posted 2011-12-19 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease; Cardiovascular Disease
Keywords: coronary artery disease; cardiovascular disease; exercise stress testing; biomarkers; NT-pro-BNP
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this study is to examine whether changes in biomarkers during exercise are related to coronary artery disease demonstrated by coronary angiography or echocardiography.

DETAILED DESCRIPTION:
Chest pain/discomfort is a common patient complaint in patients referred to outpatient clinics and emergency departments. The initial goal of evaluation is to exclude potential life threatening conditions like coronary artery disease. Exercise stress testing is a widely available non-invasive test in patients with chest pain and suspected coronary artery disease. However, the sensitivity and specificity of the test is relatively low. Exercise seems to cause an increase in the secretion of B-type natriuretic peptide (BNP), and myocardial ischemia may lead to an even more pronounced increase. Investigators aim to examine whether changes in bloodborne biomarkers such as NT-pro-BNP during exercise may improve the accuracy of exercise stress testing in patients with chest pain/discomfort and a clinical suspicion of coronary artery disease. Also, investigators aim to examine whether changes in biomarkers during exercise are related to cardiac disease demonstrated by echocardiography.

It is known that sudden heavy physical load can trigger myocardial infarction, especially in untrained individuals. The underlying mechanisms are poorly understood and may partly be related to changes in inflammation and haemostasis in patients with coronary artery disease. By measuring markers of inflammation and haemostasis during exercise stress testing, investigators hope to gain new insights into mechanisms responsible for exercise-related myocardial infarction.

Investigators also aim to do a follow-up study to investigate whether results of the initial examinations can relate to future risk of cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion criteria

* Patients referred to Oslo University Hospital Ullevål with chest pain/discomfort of unknown etiology and and a clinical suspicion of coronary artery disease.
* Intermediate or high pre test probability of coronary artery disease.
* Able to give informed, written consent.

Exclusion criteria

* Not able to perform the exercise test.
* Evidence of acute coronary syndrome.
* Known coronary artery stenosis where exercise testing is contraindicated.
* The presence of known moderate to severe valvular heart disease.
* Known heart failure or obvious clinical signs of heart failure.
* Ongoing atrial fibrillation or atrial flutter.
* Complete or partial bundle branch block.
* Digitoxin therapy.
* Pacemaker.
* Renal insufficiency (S-creatinine >150 micromol/L).
* Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients with chest pain/discomfort referred for exercise stress testing at Oslo University Hospital, including patients with acute chest pain referred to the emergency department, and referrals to the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2011-12; Primary Completion 2017-10 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease demonstrated by coronary angiography | baseline

SECONDARY OUTCOMES:
Future cardiovascular morbidity and mortality | Up to 29 years
  Investigators aim to do a follow-up study some years after enrollment to examine whether the results of the initial examinations can relate to future cardiovascular morbidity or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Arnljot Flaa, MD PhD, Study Chair — Oslo University Hospital; Ingebjørg Seljeflot, Professor PhD, Study Director — Oslo University Hospital and University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Hansen CH, Cwikiel J, Bratseth V, Arnesen H, Flaa A, Seljeflot I. Effect of Revascularization on Exercise-Induced Changes in Cardiac and Prothrombotic Biomarkers in Patients with Coronary Artery Disease. Clin Appl Thromb Hemost. 2022 Jan-Dec;28:10760296221094029. doi: 10.1177/10760296221094029. PMID 35437054
- [Derived] Cwikiel J, Seljeflot I, Berge E, Arnesen H, Wachtell K, Ulsaker H, Flaa A. Pro-coagulant activity during exercise testing in patients with coronary artery disease. Thromb J. 2017 Jan 19;15:3. doi: 10.1186/s12959-016-0127-8. eCollection 2017. PMID 28115916